CLINICAL TRIAL: NCT01341184
Title: A Phase I Open-Label Trial To Investigate the Pharmacokinetic Interaction Between Rifabutin Or Rifampin And A Single Dose Of TMC207 In Healthy Subjects
Brief Title: TMC207 +/- Rifabutin/Rifampin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0043; HHSN272201500007I
Record Dates: First submitted 2011-04-07; First posted 2011-04-25 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04-14

CONDITIONS: Tuberculosis
Keywords: rifabutin; rifampin; TMC207; tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Rifabutin; Rifampin; bedaquiline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): 16 subjects: TMC207 400mg orally on days 1 and 29, rifabutin 300mg orally, every day on day 20-41
  Interventions: Drug: Rifabutin; Drug: TMC207
- Group 2 (Experimental): 16 subjects: TMC207 400mg orally on days 1 and 29, rifampin 600mg orally, every day on day 20-41
  Interventions: Drug: Rifampin; Drug: TMC207

INTERVENTIONS:
Drug: Rifabutin — Rifabutin 300 mg orally on days 20-41
  Arms: Group 1
Drug: Rifampin — Rifampin 600 mg orally on days 20-41
  Arms: Group 2
Drug: TMC207 — TMC207 400 mg orally on days 1 and 29

SUMMARY:
Evaluation of effect of rifampin or rifabutin on single dose PK of TMC207 in healthy volunteers

DETAILED DESCRIPTION:
32 (16 per treatment group) healthy male or female subjects, 18 - 45 years old will be enrolled.Subjects will receive two single oral doses of 400mg TMC207, first on Study Day 1 followed by a 28-day wash-out, the second on Study Day 29. On Study Day 28, any abnormal safety labs will be reviewed by study physician and be determined not to meet the exclusion criteria before administration of the second dose of TMC207. Rifabutin 300mg (Group 1) or rifampin 600mg (Group 2) will be administered once daily during Period 2 from Study Day 20 through Study Day 41. The primary endpoint for the study (pharmacokinetics, safety and tolerability of TMC207 (and its M2 metabolite) will be determined on the final study visit, Day 57 (28 days after the last TMC207 dose in Period 2).

ELIGIBILITY:
Inclusion Criteria:

-Aged between 18 and 45 years, extremes included. -Non tobacco/nicotine using (at least 3 months prior to screening). -Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to <35.0 kg/m^2 -Informed Consent Form (ICF) signed voluntarily before the first trial-related activity. -Able to comply with protocol requirements. -Healthy on the basis of a medical evaluation or history that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, electrocardiogram (ECG), vital signs, ophthalmologic exam, the results of blood biochemistry, and hematology tests, and a urinalysis carried out at screening (See Section 7.2). -Subjects will be enrolled in this study only if they have undergone vasectomy/complete hysterectomy, tubal ligation, or other sterilizing procedure, or the subject is a post-menopausal woman for more than two years, or if sexually active subjects agree to use two of the following forms of adequate contraception during the study and for 12 weeks after the final dose: abstinence, condoms with or without spermicide gel, diaphragm with spermicide gel, hormonal or non-hormonal intrauterine device, oral contraceptive pills, and depot progesterone injections. If a subject is usually not sexually active but becomes active, the subject and his or her partner must use two of the listed contraceptive methods.

Exclusion Criteria:

Medical History -History or evidence of current use of alcohol, barbiturate, amphetamine, recreational, or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the trial procedures. -Any clinically significant (as deemed by the Principal Investigator) history of acute illness (resolved within 4 weeks of screening), asthma, or presence of cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (including eating disorders), endocrine, metabolic, immunologic, dermatologic, neurologic, psychological, or psychiatric disease. -Currently significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability. -Any history of significant skin disease such as, but not limited to, rash or eruptions, drug allergies, food allergy, dermatitis, eczema, psoriasis, or urticaria. Subjects with a history of skin disease may be enrolled into the study after consultation with the Sponsor Medical Monitor. -Previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication administered in this trial (i.e., rifabutin, rifampin, and TMC207). -Subjects with QTcB [Bazett correction] interval > 450ms at screening -Subjects with any other clinically significant Electrocardiogram (ECG) abnormality at screening, such as arrhythmia, ischemia, or evidence of heart failure or with a family history of Long QT Syndrome. -History or evidence of ophthalmologic diseases except for routine corrected hyperopia, myopia, and presbyopia. -Recent history (within past 30 days) of vertigo/nausea. Specific Treatments -Current use of any azole antifungal agent -Use of concomitant medication, including over-the-counter products and dietary supplements, without approval from study staff. Subjects will be treated based on symptom presentation, with the exception of medications that affect p450 and 3a metabolic pathways (refer to the MOP for a list of acceptable medications). During outpatient time periods, subjects will be required to discuss with the study staff and receive approval before self-administering any medication. After gaining approval, subjects will also be asked to record any medication taken during outpatient time periods in a provided log. -Participation in an investigational drug trial within 60 days prior to the first intake of trial medication and during the duration of the study. -Donation of blood or significant loss of blood within 56 days or plasma donation within 7 days preceding the first intake of trial medication. -Having received TMC207 in a previous trial. Based on Laboratory Abnormalities -Positive HIV-1 or HIV-2 test by Enzyme-linked immunosorbent assay (ELISA) at screening. -Hepatitis A, B, or C infection (confirmed by hepatitis A antibody IgM, hepatitis B surface antigen, or hepatitis C virus antibody, respectively) at screening. -A positive urine drug test at screening. Urine will be tested to check the current use of amphetamines, benzodiazepines, cocaine, cannabinoids, and opioids; along with serum alcohol level. -Subjects with the following laboratory abnormalities at screening as defined by the National Institute of Health (NIH), National Institute of Allergy and Infectious Diseases (NIAID), Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table (Appendix C) and in accordance with the normal ranges of the clinical laboratory: a.Serum creatinine grade 1 or greater [> 1.0 x Upper limit of lab normal range (ULN)], b.Pancreatic lipase grade 1 or greater (> 1.0 x ULN), c.Hemoglobin grade 1 or greater (</= 10.5 g/dL), d.Platelet count grade 1 or greater (</= 99000/mm^3), e.Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) grade 1 or greater (> 1.0 x ULN), f.Total bilirubin grade 1 or greater (> 1.0 x ULN), g.Creatine kinase grade 1 or greater (>1.0 x ULN), h.Troponin grade 1 or greater (1.0 x UNL), or i.Any other toxicity grade 2 or above, including: proteinuria (spot urine) > 1+ and gross hematuria. For the second dose of TMC207, any other toxicity grade 3 or above, including: proteinuria (spot urine) > 1+ and gross hematuria

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-10-21 (Actual); Primary Completion 2012-05-23 (Actual); Study Completion 2012-05-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profiles determined for Rifabutin + desacetyl rifabutin | Day 27-Day 30, Day 35 & Day 41
Pharmacokinetic profiles determined for Rifampin + desacetyl rifampin | Day 27-Day 30, Day 35 & Day 41
Pharmacokinetic profiles for TMC207 and M2 | Day 1 - Day 15
Pharmacokinetic profiles for TMC207 and M2 in combination with steady-state rifabutin (Group 1) | Day 29 - Day 41
Pharmacokinetic profiles for TMC207 and M2 in combination with steady-state rifampin (Group 2) | Day 29 - Day 41
Safety of TMC207 | Over 60 days
Tolerability of TMC207 | Over 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University - Case Medical Center - Infectious Disease & HIV Medicine, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Healan AM, Griffiss JM, Proskin HM, O'Riordan MA, Gray WA, Salata RA, Blumer JL. Impact of Rifabutin or Rifampin on Bedaquiline Safety, Tolerability, and Pharmacokinetics Assessed in a Randomized Clinical Trial with Healthy Adult Volunteers. Antimicrob Agents Chemother. 2017 Dec 21;62(1):e00855-17. doi: 10.1128/AAC.00855-17. Print 2018 Jan. PMID 29061739